CLINICAL TRIAL: NCT07248748
Title: Effects of Alexander Technique in Children With Upper Cross Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/SHANZACHAUDHARY
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: CHILD Syndrome
Keywords: Upper Cross Syndrome, Alexander Technique
MeSH Terms: conditions — Congenital Hemidysplasia with Ichthyosiform Erythroderma and Limb Defects; Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: This randomized clinical trial will involve 50 participants aged 13 to 16, recruited from Faisal Hospital Faisalabad and different schools nearby. Participants will be randomly assigned to either the Alexander Technique group, which will include home-based exercises supervised by parents, or a control group performing traditional posture-corrective exercises. The outcomes will be measured using tools such as the Cranio-Vertebral Angle (CVA), Shoulder Protraction Measurement (SPM), Thoracic Kyphotic Angle (TKA), and Visual Analogue Scale (VAS) for pain assessment. The findings are expected to provide insights into the benefits of the Alexander Technique as a therapeutic strategy for addressing UCS and improving overall health outcomes in adolescents. Data collection will be done before and after the intervention. Data will be analyzed through SPSS version 26.00.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Active Comparator): control group
  Interventions: Other: Corrective exercises
- GROUP B (Active Comparator): interventional group
  Interventions: Other: Alexander technique

INTERVENTIONS:
Other: Alexander technique — In the AT group, parents will supervise the patients exercises at home base on the explanations and training the corrective movements specialist provided in the first session. In the AT group, adolescents were taught the considerations and habits they should remember and focus on daily basis. These included teaching ergonomic considerations and individual postural habits during daily activities such as standing, walking, sitting, sleeping, reading, using a computer, and other repetitive and continuous activities performed during the day.
  Arms: GROUP B
Other: Corrective exercises — The Corrective exercises will be done in home base setting, and the corrective movements' specialist will be responsible for supervising their performance twice a week. Selected CE will designed to correct posture and address the mentioned abnormalities through stretching exercises for shortened muscles and strengthening exercises for individuals with weak muscles. These exercises will include a 5-10-minute warm-up followed by stretching exercises for the chest, hip- flexor-psoas, upper trapezius, intercostal muscles, upper neck extensors, and then strengthening exercises for the shoulder protractors, deep neck flexors, lower neck extensors, and thoracic spine extensors
  Arms: GROUP A

SUMMARY:
This randomized clinical trial will involve 50 participants aged 13 to 16, recruited from Faisal Hospital Faisalabad and different schools nearby. Participants will be randomly assigned to either the Alexander Technique group, which will include home-based exercises supervised by parents, or a control group performing traditional posture-corrective exercises. The outcomes will be measured using tools such as the Cranio-Vertebral Angle (CVA), Shoulder Protraction Measurement (SPM), Thoracic Kyphotic Angle (TKA), and Visual Analogue Scale (VAS) for pain assessment. The findings are expected to provide insights into the benefits of the Alexander Technique as a therapeutic strategy for addressing UCS and improving overall health outcomes in adolescents. Data collection will be done before and after the intervention. Data will be analyzed through SPSS version 26.00.

DETAILED DESCRIPTION:
Upper Cross Syndrome (UCS) is a common postural disorder characterized by muscle imbalances resulting from prolonged use of electronic devices, leading to symptoms such as forward head posture, rounded shoulders, and increased thoracic kyphosis. This condition predominantly affects young adults and is associated with discomfort and decreased postural stability, negatively impacting overall physical function. The study aims to investigate the effectiveness of the Alexander Technique (AT) in improving pain levels and range of motion (ROM) in individuals with Upper Cross Syndrome. By focusing on the principles of optimal body use and postural awareness, the Alexander Technique may offer a valuable intervention to alleviate symptoms and enhance Range of motion.

This randomized clinical trial will involve 50 participants aged 13 to 16, recruited from Faisal Hospital Faisalabad and different schools nearby. Participants will be randomly assigned to either the Alexander Technique group, which will include home-based exercises supervised by parents, or a control group performing traditional posture-corrective exercises. The outcomes will be measured using tools such as the Cranio-Vertebral Angle (CVA), Shoulder Protraction Measurement (SPM), Thoracic Kyphotic Angle (TKA), and Visual Analogue Scale (VAS) for pain assessment. The findings are expected to provide insights into the benefits of the Alexander Technique as a therapeutic strategy for addressing UCS and improving overall health outcomes in adolescents. Data collection will be done before and after the intervention. Data will be analyzed through SPSS version 26.00.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13 -16
* School going children

Exclusion Criteria:

* Participants with signs of:
* Fractures
* Surgeries
* Joint problems
* Injuries in the spine
* Skeletal-muscular imbalances
* Lower limb cross syndrome abnormal BMI participants engaging in regular physical activity for at least 6 h per week

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Cranio-vertebral angle (CVA) | 8 weeks
  Cranio-vertebral angle (CVA) is the most widely known measurement method used to determine how forward the head is tilted in a person in FHP. For CVA measurement, the digital camera (Canon 650D, Canon, Japan) was fixed and mounted at a distance of 1m, and the side of the subject was photographed, for accurate measurement of CVA, a plumb line suspended from the ceiling was allowed to descend directly next to the subject.Subjects were instructed to stand comfortably with both arms relaxed on the side of the trunk and maintain a natural head posture.
  CVA was defined as the angle between the horizontal line and the line from the spinous process of the seventh cervical vertebra to the ear tragus. The CV angle means that the smaller the angle, the greater the flexion of the lower cervical spine
Shoulder Protraction Measurement (SPM) | 8 weeks
  The complexity of these combined motions as well as the thick surrounding soft tissues present challenges to accurate angular measurement of scapular motion. However, observing these scapular motions superiorly provides a perspective of the superficial acromion as an indicator of scapular position relative to the medial superior angle and therein may lie the opportunity for goniometric assessment.
Thoracic Kyphotic Angle (TKA) | 8 weeks
  The thoracic kyphotic angle (TKA) is defined as the angle formed by the intersection of two lines drawn along the superior endplate of the uppermost thoracic vertebra and the inferior endplate of the lowermost thoracic vertebra. This angle is crucial for assessing spinal alignment and postural abnormalities.
Visual Analogue Scale (VAS) | 8 weeks
  VAS is widely used as a measure of pain intensity in globally. It has been shown that VAS is valid, reliable and interval scale. VAS has high testretest reliability and repeatability. In this VAS, it has a continuous scale consist of a horizontal and vertical line that called vertical VAS and horizontal visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shanza Chaudhary, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Asif Javed, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Neill MM, Anderson DI, Allen DD, Ross C, Hamel KA. Effects of Alexander Technique training experience on gait behavior in older adults. J Bodyw Mov Ther. 2015 Jul;19(3):473-81. doi: 10.1016/j.jbmt.2014.12.006. Epub 2015 Jan 7. PMID 26118520